CLINICAL TRIAL: NCT03340857
Title: Evaluation of the Use of an Intelligent Electric Bicycle for Health (VELIS) to Optimize the Return to Physical Activity After a Stay for Effort Retraining in Rehabilitation and Recuperative Care Facilities for Oncology Patients
Brief Title: Intelligent Electric Bicycle for Health (VELIS) to Optimize the Return to Physical Activity for Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Audavie (Other)
Collaborators: Floralis (Industry); eBikeLabs (Unknown); Rocheplane Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ONCOVELIS version 2.0
Record Dates: First submitted 2017-09-27; First posted 2017-11-14 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Cancer; Oncology
Keywords: Post-cancer retraining; Physical activity; Intelligent electric bicycle
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intelligent electric bicycle (VELIS) sessions (Experimental): Intelligent electric bicycle (VELIS) sessions with an instructor, twice a week for 6 weeks
  Interventions: Other: Intelligent electric bicycle (VELIS) sessions

INTERVENTIONS:
Other: Intelligent electric bicycle (VELIS) sessions — Oncology patients will participate in intelligent electric bicycle (VELIS) sessions twice a week for 6 weeks after their release from a rehabilitation and recuperative care facility

SUMMARY:
The purpose of this pilot study is to encourage oncology patients to continue effort retraining after their release from rehabilitation and recuperative care facilities with physical activity sessions and therapeutic education using an intelligent electric bicycle (VELIS)

DETAILED DESCRIPTION:
The benefit of physical activity in oncology is now clearly established. Physical activity has its place at all stages of the fight against cancer in primary, secondary and tertiary prevention.

Rehabilitation and recuperative care facilities may be a first step for patients with significant deconditioning, but long-term benefits are essential.

Nevertheless, the post rehabilitation and recuperative care facilities transition period is for these patients a temporary period during which they may loose part of the benefit of effort retraining and physical reconditioning.

The investigators believe that it is necessary to go beyond the "physiological" efficiency to identify and overcome the patient's stereotypes regarding physical activity, to customize and adapt the programs to each patient, and to bring quickly the notion of pleasure and success in the practice of physical activity. Electrically assisted bicycles can reach most of these goals provided that they are adapted.

The objective of this project is to set up and evaluate, thanks to a monocentric pilot study, a process of continuation of exercise retraining through physical activity and therapeutic education sessions for the promotion of physical activity, focusing on the use of electrically assisted bicycles, in continuation of an exercise retraining in rehabilitation and recuperative care facilities.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over
* Patient who has followed a post-cancer effort retraining program in a rehabilitation facility at Rocheplane Medical Center
* Patient with the ability to pedal on an outdoor bicycle
* Patient with no restriction to moderate physical activity or bicycling (acute coronary disease of less than 2 years, locomotor problem of the spine or lower limbs incompatible with the practice of cycling)
* Weight less than 125 kg (maximum load for VELIS)
* Patient available for a 4 months follow-up

Exclusion Criteria:

* Patient with a restriction to the practice of moderate physical activity or bicycle (acute coronary disease of less than 2 years, locomotor problem)
* Persons referred to in Articles L1121-5 to L1121-8 of the CSP (corresponds to all protected persons), pregnant, parturient, nursing mother, person deprived of liberty by judicial or administrative decision, a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reaching the goal of 150 min equivalent of moderate physical activity per week (600 MET-min/week) | 4 Months
  Evaluated with the IPAQ questionnaire short version (International Physical Activity Questionnaire)

SECONDARY OUTCOMES:
Quantitative analysis of kinetic physical activity evolution | Enrollment and then once a month from Month 2 to Month 4, the last week of the month, velis sessions and effort retraining excluded
  Longitudinal continue quantitative data from IPAQ score
Evaluate the VELIS sessions feasibility n°1 | 4 Months
  Number of cancelled sessions
Evaluate the VELIS sessions feasibility n°2 | 4 Months
  Number of incomplete sessions
Evaluate the VELIS sessions feasibility n°3 | 4 Months
  Collection of the failure reasons by the instructor
Evaluate the impact on the physical capacities n°1 | 4 Months
  Progression of the patients physical activity (clinical exam weight)
Evaluate the impact on the physical capacities n°2 | 4 Months
  Progression of the patients physical activity (heart rate)
Evaluate the impact on the physical capacities n°3 | 4 Months
  Progression of the patients physical activity (analysis of physio-cardiological criteria)
Evaluate the impact on the physical capacities n°4 | 4 Months
  Analysis of the progression during intelligent electric bicycle (VELIS) sessions with associated factors (initial gain in effort retraining)
Evaluate the impact on the physical capacities n°5 | 4 Months
  Analysis of the progression during intelligent electric bicycle (VELIS) sessions with associated factors (age)
Evaluate the impact on the physical capacities n°6 | 4 Months
  Analysis of the progression during intelligent electric bicycle (VELIS) sessions with associated factors (gender)
Evaluate the impact on the physical capacities n°7 | 4 Months
  Analysis of the progression during intelligent electric bicycle (VELIS) sessions with associated factors (pathologies)
Evaluate the impact on the physical capacities n°8 | 4 Months
  Constant-Load Exercise Test at 80% MAP (Maximum Aerobic Power) (endurance test on ergocycle)
Evaluate the impact on the physical capacities n°9 | 4 Months
  Constant-Load Exercise Test at 80% MAP (Maximum Aerobic Power) (evaluation with the quantitative Borg scale (from Pr Gunnar BORG) from 0 to 10 (the goal score is 4 to 5)).
Evaluate the impact on the physical capacities n°10 | 4 Months
  Constant-Load Exercise Test at 80% MAP (Maximum Aerobic Power) (heart rate)
Evaluate the impact on the physical capacities n°11 | 4 Months
  Constant-Load Exercise Test at 80% MAP (Maximum Aerobic Power) (visual analogical scale from 0 (no pain) to 10 (maximal pain) for the lower limbs pain. Lower value is a better outcome)
Evaluate the impact on the physical capacities n°12 | 4 Months
  Measurement of the muscular power using a handgrip (physiological parameter). Higher value is a better outcome.
Improve quality of life | 4 Months
  Euroquol 5 dimensions scale (from 0 to 100 : higher value is a better outcome)
Improve fatigue n°1 | 4 Months
  Analogic visual scale about fatigue once a month
Improve fatigue n°2 | 4 Months
  Fatigue Piper score
Improve chronic pain | 4 Months
  Analogic visual scale about pain once a month
Improve self-esteem | 4 Months
  Evaluation with Rosenberg score
Improve patient satisfaction | 4 Months
  Satisfaction survey and wish to do again intelligent electric bicycle (VELIS) sessions or to continue electric bicycle sessions
Remove stereotypes that can lead to inhibition in the physical activity practice | 4 Months
  Evaluation of the psychological representation of physical activity using the Cancer Exercise Stereotypes Scale (CESS) questionnaire from the SENS (sport and social environment laboratory) team from Grenoble.
  The average value is calculated for each subscale.
  Adherence to positive stereotypes if value is below 4 for the following subscale :
  * Lack of interest in physical activity (items 1, 6, 11)
  * Side effects related to treatment (items 3, 8, 13, 17)
  * Risks related to physical activity (items 5, 10, 15) Adherence to positive stereotypes if value is greater than 4 for the subscale Benefits of physical activity (items 4, 9, 14, 18).
Evolution of uses and performances during bicycle sessions at the beginning and the end of the intervention n°1 | 6 weeks
  Analysis of the parameters profiles recorded by the VELIS : heart rate monitor
Evolution of uses and performances during bicycle sessions at the beginning and the end of the intervention n°2 | 6 weeks
  Analysis of the parameters profiles recorded by the VELIS : speed
Evolution of uses and performances during bicycle sessions at the beginning and the end of the intervention n°3 | 6 weeks
  Analysis of the parameters profiles recorded by the VELIS : electric power provided by the engine
Evolution of uses and performances during bicycle sessions at the beginning and the end of the intervention n°4 | 6 weeks
  Analysis of the parameters profiles recorded by the VELIS : rate of pedaling for the reference itinerary

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Bosson, MD, Principal Investigator — Laboratoire TIMC - Themas
Locations (1):
- Rocheplane Medical Center, Saint-Martin-d'Hères, Auvergne-Rhône-Alpes, France

REFERENCES:
- [Background] Phillips SM, Alfano CM, Perna FM, Glasgow RE. Accelerating translation of physical activity and cancer survivorship research into practice: recommendations for a more integrated and collaborative approach. Cancer Epidemiol Biomarkers Prev. 2014 May;23(5):687-99. doi: 10.1158/1055-9965.EPI-13-1355. Epub 2014 Mar 5. PMID 24599577
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A; American College of Sports Medicine; American Heart Association. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1081-93. doi: 10.1161/CIRCULATIONAHA.107.185649. Epub 2007 Aug 1. PMID 17671237
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1435-45. doi: 10.1249/mss.0b013e3180616aa2. PMID 17762378
- [Background] Mielgo-Ayuso J, Aparicio-Ugarriza R, Castillo A, Ruiz E, Avila JM, Aranceta-Batrina J, Gil A, Ortega RM, Serra-Majem L, Varela-Moreiras G, Gonzalez-Gross M. Physical Activity Patterns of the Spanish Population Are Mostly Determined by Sex and Age: Findings in the ANIBES Study. PLoS One. 2016 Feb 25;11(2):e0149969. doi: 10.1371/journal.pone.0149969. eCollection 2016. PMID 26914609
- [Background] Pavey TG, Anokye N, Taylor AH, Trueman P, Moxham T, Fox KR, Hillsdon M, Green C, Campbell JL, Foster C, Mutrie N, Searle J, Taylor RS. The clinical effectiveness and cost-effectiveness of exercise referral schemes: a systematic review and economic evaluation. Health Technol Assess. 2011 Dec;15(44):i-xii, 1-254. doi: 10.3310/hta15440. PMID 22182828
- [Background] Welker J, Cornuz J, Gojanovic B. [Electrically assisted bicycles: health enhancement or "green" gadget?]. Rev Med Suisse. 2012 Jul 25;8(349):1513-7. French. PMID 22913003
- [Background] Peterman JE, Morris KL, Kram R, Byrnes WC. Pedelecs as a physically active transportation mode. Eur J Appl Physiol. 2016 Aug;116(8):1565-73. doi: 10.1007/s00421-016-3408-9. Epub 2016 Jun 14. PMID 27299435
- [Background] Gojanovic B, Welker J, Iglesias K, Daucourt C, Gremion G. Electric bicycles as a new active transportation modality to promote health. Med Sci Sports Exerc. 2011 Nov;43(11):2204-10. doi: 10.1249/MSS.0b013e31821cbdc8. PMID 22005715
- [Background] Simons M, Van Es E, Hendriksen I. Electrically assisted cycling: a new mode for meeting physical activity guidelines? Med Sci Sports Exerc. 2009 Nov;41(11):2097-102. doi: 10.1249/MSS.0b013e3181a6aaa4. PMID 19812505
- [Background] Falzon C, Sabiston C, Bergamaschi A, Corrion K, Chalabaev A, D'Arripe-Longueville F. Development and validation of the Cancer Exercise Stereotypes Scale. J Psychosoc Oncol. 2014;32(6):708-26. doi: 10.1080/07347332.2014.955237. PMID 25174265
- [Background] Piper BF, Dibble SL, Dodd MJ, Weiss MC, Slaughter RE, Paul SM. The revised Piper Fatigue Scale: psychometric evaluation in women with breast cancer. Oncol Nurs Forum. 1998 May;25(4):677-84. PMID 9599351
- See also: 3rd report INCA february 2017 — http://www.e-cancer.fr/Expertises-et-publications/Catalogue-des-publications/Troisieme-rapport-au-president-de-la-Republique-Fevrier-2017
- See also: Evaluation of the impact on health. Promotion of the electrical bike. Final report. 2006 — http://www.impactsante.ch/pdf/EIS_VAE_2006.pdf
- See also: Gretchen Reynolds. The Surprising Health Benefits of an Electric Bike JULY 6, 2016 6:00 AM July 6, 2016. — http://well.blogs.nytimes.com/2016/07/06/the-surprising-health-benefits-of-an-electric-bike-2/?smid=tw-nytimes&smtyp=cur&_r=1